CLINICAL TRIAL: NCT07348705
Title: Electrophysiology-based Deep Brain Stimulation Programming for Parkinson's Disease
Brief Title: Electrophysiology-based DBS Programming for PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202500821
Record Dates: First submitted 2026-01-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD)
Keywords: deep brain stimulation; DBS; PD; Parkinson's disease; beta power
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Clinician-based (Active Comparator)
  Interventions: Device: Clinician-based DBS programming
- Maximum beta power-based (Active Comparator)
  Interventions: Device: Maximum Beta power-based DBS programming
- Broad-band (Experimental)
  Interventions: Device: Broad-band electrophysiology-based DBS programming

INTERVENTIONS:
Device: Clinician-based DBS programming — Contacts, amplitude, pulse width, and frequency are chosen by the treating physician during a conventional monopolar review.
  Arms: Clinician-based
Device: Maximum Beta power-based DBS programming — The contact that shows the strongest beta activity (13-30 Hz) in the local field potentials is selected for stimulation.
  Arms: Maximum beta power-based
Device: Broad-band electrophysiology-based DBS programming — A multi-frequency algorithm that integrates beta, theta/alpha, finely tuned gamma, and other relevant bands is used to identify the optimal contact.
  Arms: Broad-band

SUMMARY:
Deep brain stimulation (DBS) effectively alleviates motor symptoms in Parkinson's disease (PD). However, current programming is manual and time-consuming. This study will evaluate physiology-based programming using local field potentials (LFPs) to identify optimal stimulation parameters. Specifically, DBS contact selection based on beta power and a broad-band approach will be compared with conventional clinician-based programming.

DETAILED DESCRIPTION:
Up to thirty patients with DBS (unilateral or bilateral leads) attached to a bidirectional implantable pulse generator will be enrolled in this study. This commercially available IPG allows both therapeutic stimulation and chronic sensing. It has been designed to capture local field potentials (LFPs) from implanted DBS leads while delivering stimulation both inside and outside the clinic.

After recording LFP data, then, the physician will perform the traditional clinical monopolar review and determine the optimized DBS settings ('clinician-based' settings) following standard clinical procedures, and without looking at the physiology data. In parallel, the LFP data will be analyzed to identify the 'optimal' therapy contact based on 1) maximum beta power, and 2 ) broad-band multi-frequency analysis.

The physician will then setup up to 4 stimulation programs will be set up:

1. Clinician-based programming (standard of care),
2. Maximum Beta power-based programming,
3. Broad-band programming.
4. If needed, second-best clinician-based programming (standard of care)

In this study, settings 1, 2, and 4 (optional) are determined based on established standards of care or manufacturer guidelines. Setting 3, however, is derived using our novel electrophysiology-based algorithm. While the method for determining this setting is innovative, the resulting parameter may be identical to those obtained through conventional approaches (settings 1, 2, or 4). Therefore, although the methodology introduces a new process, the final settings remain within clinically accepted ranges and do not exceed standard clinician-based practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of idiopathic PD fulfilling the Movement Disorder Society Clinical Diagnostic Criteria for PD
* DBS implantation with the Percept DBS device (Medtronic, USA) for the treatment of motor symptoms
* Ability to give informed consent for the study
* Willingness to do this study at the time of the initial programming session
* Age 21 to 89 years old

Exclusion Criteria:

* Inability to comply with the study protocol
* Atypical Parkinsonism
* Any personality or mood symptoms that study personnel believe will interfere with the study requirements

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2031-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of motor symptoms using the Unified Parkinson's Disease Rating Scale (UPDRS) | From enrollment to end of study (1 month)
  The UPDRS (Unified Parkinson's Disease Rating Scale) Motor Scale (Part III) is a clinician-rated tool assessing motor functions like tremor, rigidity, bradykinesia, and gait in Parkinson's disease (PD), using a 0-4 scale for each item, with higher scores indicating greater impairment, helping track disease progression and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wong, MD, Principal Investigator — University of Florida
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States